CLINICAL TRIAL: NCT04640857
Title: Randomized Double Blind Controlled Prospective Study to Evaluate the Influence of Radiofrequency Based Toothbrush on the Accumulation of the Calculus
Brief Title: Evaluation of the Influence of Radiofrequency-based Toothbrush on the Accumulation of Calculus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0352-20-RMB CTIL
Record Dates: First submitted 2020-11-01; First posted 2020-11-23 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Oral Hygiene
Keywords: Electromagnetic Fields; Oral Hygiene

STUDY DESIGN:
Intervention Model Description: Experimental: Silk'n Toothwave
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group: Silk'n Toothwave with vibration and electromagnetic field (Experimental): Silk'n Toothwave with vibration and electromagnetic field use twice a day for 3 months.
  Interventions: Device: Silk'n Toothwave
- Control group: Silk'n Toothwave with-out an electromagnetic field ( only vibration) (Sham Comparator): Silk'n Toothwave without an electromagnetic field (only vibration ) use twice a day for 3 months.
  Interventions: Device: Silk'n Toothwave
- Silk'n Toothwave with an electromagnetic field and without vibration (Active Comparator): Silk'n Toothwave with an electromagnetic field and without vibration use twice a day for 3 months.
  Interventions: Device: Silk'n Toothwave

INTERVENTIONS:
Device: Silk'n Toothwave — patients will receive a non-surgical treatment which will include oral hygiene instructions, calculus removal with ultrasonic and manual instruments. At the end of the meeting they will be provided with a toothbrush which is based on a radiofrequency technology.

SUMMARY:
to evaluate the influence of radiofrequency based toothbrush (Silk'n toothwave)on the accumulation of the calculus

DETAILED DESCRIPTION:
Calculus is a white-brownish layer with various levels of stiffness, which accumulates on teeth and is formed by the mineralization of dental plaque.

Thus, maintaining oral hygiene and adhering to maintenance programs keep low levels of plaque and calculus.

The electromagnetic field is known for bone healing by lessening osteoclast activity, improving osteoid formation, and stimulating angiogenesis. Furthermore, the electromagnetic field has an antimicrobial effect.

Electric toothbrushes have shown a statistical reduction in plaque accumulation and gingival inflammation.

Previous studies have shown that Silk'n Toothwave results in less plaque accumulation and calculus formation, in addition to stain removal and teeth whitening.

Study aim: to asses the effect of the electromagnetic field in a tooth brush (Silk'n Toothwave) on calculus accumulation and gingival parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 20-85 Years old
* Subject must have voluntarily signed the informed consent form before any study related action
* Presence of gingival inflammation (Gingival Index by Silness and Loe 1969)
* Presence of plaque on clinical crowns (calculation of area)
* Supportive periodontal therapy (with ultra-sonic and manual devices) on a regular basis with a 3-month interval with a minimum of 3 times in a row prior to T0 (baseline)
* Compliance with study schedules and arrival at study visits

Exclusion Criteria:

* A systemic or pharmacological condition that can affect the healing of soft or hard tissue in the rest of the teeth or implants such as cyclosporine, calcium channel blockers
* Pregnant or lactating women (*If Male Please write N/A).
* Heavy smokers (more than 10 cigarettes per day).
* Patients with a pacemaker that do not allow the use of an ultrasonic device.
* Patient with an active periodontal disease (may undergo periodontal treatment as required and not completed as part of the study if it can be included in the study).
* Systemic condition requiring prophylactic antibiotics.
* Patients taking NSAIDS for prolonged period.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Plaque score % | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  to estimate the presence of plaque and its accumulation on the tooth surface of anterior mandibular incisors
Change in Calculus ratio % | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  to estimate the percentage of calculus on the lingual aspect of anterior mandibular incisors using ImageJ software
Change in Free gingival margin color (CEILAB color space) | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  the color of the gingiva will be measured with the software Adobe photoshop and will be calculated with CIELAB color space.

SECONDARY OUTCOMES:
Probing depth mm | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  to measure the pocket depths around the anterior mandibular incisors
Bleeding on probing Yes/No | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  to document the presence or absence of bleeding of the dental pocket after probing
Recession mm | baseline (T0), after 4 weeks (T1), after 12 weeks (Tf)
  to measure the discrepancy (if existent) between the cementoenamel junction and the free gingival margin in the buccal aspect of the anterior mandibular incisors
Subject satisfaction questionnaire | 4 weeks (T1), after 12 weeks (Tf)
  the questionnaire includes 4 questions: satisfaction, convenience, improvement in oral hygiene and the quality of brushing

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Zigdon, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel

REFERENCES:
- [Derived] Khoury J, Giladi HZ, Ginesin O, Gabay E, Mayer Y. The influence of radio frequency-based toothbrush on the accumulation of calculus and periodontal health: A randomized double-blind controlled prospective study. Clin Exp Dent Res. 2023 Aug;9(4):574-585. doi: 10.1002/cre2.770. Epub 2023 Jul 29. PMID 37515446